CLINICAL TRIAL: NCT04543240
Title: The Relationship Between Bacterial Load and the Clinical Outcomes for Integra™ in Operative Wounds
Brief Title: Bacterial Load for Integra™ in Operative Wounds
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Principal Investigator, Christopher Attinger, M.D., Professor and Director of the Center for Wound Healing, Georgetown University
Other Study IDs: 2017-0908
Record Dates: First submitted 2020-09-01; First posted 2020-09-10 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Wounds and Injuries
Keywords: Lower extremity
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Integra™ dermal regeneration template — Integra a biologic dressing for deep wounds or large soft tissue defects that penetrate to the level of bone

SUMMARY:
Proportion of postoperative complications (infections, dehiscence, graft slough) after initial application of Integra™

DETAILED DESCRIPTION:
This is a study examining the use of Integra™ for the treatment of lower extremity wounds to better understand the relationship between bacteria contamination levels and post-operative complications. Wounds requiring operative application of Integra™ alone or Integra™ followed by a planned subsequent application of a STSG will be enrolled into this study.

The tolerance of Integra™ to bacterial bioburden at the time of application will be determined by observing their respective postoperative wound complications and correlating these findings with quantitative bacterial counts, qualitative culture results, and bacterial and wound protease levels at the time of Integra™ alone application or Integra™ followed by STSG application.

Patients will then be followed until complete healing has occurred or until 16 weeks, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18-90.
* Full-thickness wounds below the knee.
* Patients who require, in the opinion of the Investigator, operative application of Integra™.
* Patients able and willing to comply with the study protocol.

Exclusion Criteria:

* Male or Female under 18 or over 90
* Patients that do not have Full-thickness wounds below the knee
* Patients who do not require, in the opinion of the Investigator, operative application of Integra™.
* Patients that are not able or willing to comply with the study protocol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be anyone who is experiencing partial or full thickness wounds, pressure ulcers, venous and diabetic ulcers, burns, and traumatic wounds.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Determine a threshold in which Integra is tolerant to bacteria that yields positive results (healing). The investigators believe that this device is more tolerant to bacterial load then current perception. | 1 year
  Quantitative CFUs will be obtained by obtaining tissue from the wound at the time of debridement from otherwise discarded tissue. After tissue cultures are obtained and sent to a designated microbial lab for analysis. Tissue culture is to be obtained from the central aspect of the wound bed. These cultures will be processed and analyzed for research purposes. Qualitative cultures will be obtained as per SOC and sent to the local lab per customary fashion.
  Qualitative bacterial protease and human inflammation protease indications will be obtained by sampling and testing two separate wound fluid swabs on investigational devices; WOUNDCHEKTM Bacterial Status and WOUNDCHEKTM Protease Status. Bacterial Status detects enzymes that are present when bacteria have become pathogenic while Protease Status detects enzymes present when the wound is in a chronically inflamed state. The tests will be obtained from Woundchek Labs.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Attinger, MD, Principal Investigator — MedStar Georgetown University Hopsital
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No